CLINICAL TRIAL: NCT05485792
Title: A Prospective Study on Comparison 18F-FAPI and 18F-FDG PET/CT in the Evaluation of Patients With Various Types of Cancer
Brief Title: 18F-FAPI and 18F-FDG PET/CT in Patients With Various Types of Cancer
Acronym: FAPI-VTC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPI-malignancy
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects with various types of cancer undergo contemporaneous 18F-FAPI and 18F-FDG PET/CT either for an initial assessment or for recurrence detection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FAPI PET/CT (Experimental): Each subject undergone both 18F-FDG and 68Ga-FAPI PET/CT scans within 2 week
  Interventions: Diagnostic Test: 18F-FAPI PET/CT and 18F-FDG PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-FAPI PET/CT and 18F-FDG PET/CT — Each subject undergo both 18F-FDG and 68Ga-FAPI PET/CT scans within 1 week

SUMMARY:
FAP is overexpressed in the cancer-associated fibroblasts (CAFs) of 90% epithelial carcinomas. Currently, 68Ga-fibroblast activation protein inhibitor (FAPI) has shown promising diagnostic value in many types of tumors. However, there are currently no studies on head-to-head comparison of diagnosis value of various types of cancer in 18F-FAPI and 18F-FDG PET/CT. Therefore, we conducted a prospective study to investigate the value of 18F-FAPI PET/CT in various types of cancer, and compare it with 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Fibroblast activation protein (FAP) is a serine protease that belongs to the dipeptidyl peptidase-IV (DPP-IV) family located in fibroblast membranes. FAP is overexpressed in the cancer-associated fibroblasts (CAFs) of 90% epithelial carcinomas, including primary and metastatic liver cancer. Therefore, FAP-targeted radiopharmaceuticals can be considered a promising approach for the visualization of CAFs. CAFs are crucial component of tumor stroma, promote the growth of cancer cells and are associated with poor prognosis. Currently, Gallium 68 (68Ga)-fibroblast activation protein inhibitor (FAPI) has shown promising diagnostic value in many types of tumors, including lung cancer, gastric carcinomas, peritoneal carcinomas. However, there are currently no studies on head-to-head comparison of diagnosis value of various types of cancer in 18F-FAPI and 18F-FDG PET/CT. Therefore, we conducted a prospective study to investigate the value of 18F-FAPI PET/CT in various types of cancer, and compare it with 18F-FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (aged 18 years or order);
2. patients with suspected or newly diagnosed or previously treated malignant tumors (supporting evidence may include CT, MRI and pathology report);
3. patients who had scheduled both 18F-FAPI PET/CT and 18F-FDG PET/CT scans;
4. patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

1. patients with non-malignant lesions;
2. patients with pregnancy;
3. the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum standardized uptake value (SUVmax) | 30 days
  The SUVmax of 18F-FDG PET/CT and 18F-FAPI PET/CT

SECONDARY OUTCOMES:
The target-to-background ratio (TBR) | 30 days
  The target-to-background ratio (TBR) was calculated by dividing the SUVmax of the lesion by the SUVmax of soft tissue background

CONTACTS AND LOCATIONS:
Overall Officials: Rusen Zhang, MD, Study Director — Affiliated Cancer Hospital & Institute of Guangzhou Medical University

REFERENCES:
- [Derived] Liang J, Weng S, Zhang J, Jiang S, Li W, Li S, Rong J, Liu H, Chen H, Liu Z, Peng H, Yan S, Zhang R, Liang SH, Zhang L. Diagnostic performance of [18F]FAPI-04 PET/CT in suspected recurrent hepatocellular carcinoma: prospective comparison with contrast-enhanced CT/MRI. Eur J Nucl Med Mol Imaging. 2025 Sep;52(11):3951-3962. doi: 10.1007/s00259-025-07273-4. Epub 2025 Apr 15. PMID 40232335
- [Derived] Liang Z, Peng H, Li W, Liu Z. Head-to-head study of [18F]FAPI-04 PET/CT and [18F]FDG PET/CT for non-invasive assessment of liver cancer and its immunohistochemical markers. BMC Cancer. 2024 Nov 11;24(1):1378. doi: 10.1186/s12885-024-13153-1. PMID 39528951
- [Derived] Liang J, Jiang S, Song J, Chen D, Weng S, Li S, Peng H, Liu Z, Zhang J, Chen Y, Rao S, Chen H, Zhang R, Liu H, Zhang L. Role of [18F]FAPI-04 in staging and therapeutic management of intrahepatic cholangiocarcinoma: prospective comparison with [18F]FDG PET/CT. EJNMMI Res. 2024 Sep 11;14(1):81. doi: 10.1186/s13550-024-01145-y. PMID 39256297
- [Derived] Zhang J, Jiang S, Li M, Xue H, Zhong X, Li S, Peng H, Liang J, Liu Z, Rao S, Chen H, Cao Z, Gong Y, Chen G, Zhang R, Zhang L. Head-to-head comparison of 18F-FAPI and 18F-FDG PET/CT in staging and therapeutic management of hepatocellular carcinoma. Cancer Imaging. 2023 Oct 30;23(1):106. doi: 10.1186/s40644-023-00626-y. PMID 37899452